CLINICAL TRIAL: NCT01257919
Title: Investigator-blinded, Randomized, Cross-over, Multiple Dose Phase I Study on Safety and Pharmacokinetics of Topically Applied Azelaic Acid Foam, 15% Compared to Azelaic Acid Gel, 15% in Subjects With Papulopustular Rosacea
Brief Title: Safety and Pharmacokinetics of Azelaic Acid Foam, 15% in Papulopustular Rosacea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15386; 1401843 (Other: Company Internal)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2014-02

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic Acid Foam 15% (Experimental): Dermal application of Azelaic Acid Foam 15%
  Interventions: Drug: Azelaic Acid Foam
- Azelaic Acid Gel 15% (Active Comparator): Dermal application of Azelaic Acid Gel 15%
  Interventions: Drug: Azelaic Acid Gel

INTERVENTIONS:
Drug: Azelaic Acid Foam — Dermal application of Azelaic Acid Foam
  Arms: Azelaic Acid Foam 15%
Drug: Azelaic Acid Gel — Dermal application of Azelaic Acid Gel
  Arms: Azelaic Acid Gel 15%

SUMMARY:
Assessment of pharmacokinetics of Azelaic Acid Foam after repeated skin application and in comparison to Azelaic Acid gel.

Assessment of safety after repeated skin application.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate papulopustular rosacea
* free of any clinically significant disease

Exclusion Criteria:

* body weight less than 50 or more than 130 kg
* clinically significant disease which could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Baseline corrected area under the curve (AUC) | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Novum Pharmaceutical Research Services of Nevada Inc., Las Vegas, Nevada, United States